CLINICAL TRIAL: NCT00616109
Title: Phase II Trial of Sunitinib (Sutent, SU11248) Maintenance Therapy After Induction Platinum-Based Chemotherapy in Patients With Extensive-Stage Small Cell Lung Cancer
Brief Title: Sunitinib Maintenance Therapy After Induction Platinum-Based Chemotherapy in Patients With ES-SCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Principal Investigator, Gregory Kalemkerian. M.D., Professor of Internal Medicine, University of Michigan Rogel Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2007.034; HUM12046 (Other: IRBMED (University of Michigan Medical School IRB))
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Extensive-Stage Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Maintenance Sunitinib (Experimental): Main interventional arm of study. Subjects who received maintenance sunitinib experimentally on this study were from a population of (consenting) patients with histologically or cytologically documented Extensive-State Small Cell Lung Cancer (ES-SCLC) who did not progress (were classified as Complete Response or "CR", Partial Response or "PR", or Stable Disease or "SD") after an induction chemotherapy (Cisplatin and etoposide)
  Interventions: Drug: sunitinib

INTERVENTIONS:
Drug: sunitinib — Sunitinib will be given at 50 mg/day as a single agent for 4 consecutive weeks followed by a 2-week rest period to form a complete cycle of 6 weeks.
  Other Names: Sutent

SUMMARY:
The goal of this study is to determine the progression-free survival rate in patients with extensive-stage small cell lung cancer who had achieved complete response, partial response, or stable disease with their previous platinum chemotherapy regimen, such as cisplatin or carboplatin in combination with etoposide or irinotecan. In addition, the safety and effectiveness of sunitinib will also be evaluated.

DETAILED DESCRIPTION:
Despite a high initial response rate, all patients with extensive-stage small cell lung cancer treated with standard chemotherapy will develop disease progression, usually within one year of initial treatment. Therefore, prolonging progression-free survival in this disease is meaningful for clinical trials exploring agents such as sunitinib. Sunitinib is a drug that inhibits the biological pathway responsible for the growth and spread of cancer cells. For this reason, we believe that sunitinib maintenance therapy will delay or prevent recurrence and prolong survival.

The goal of this study is to determine the progression-free survival rate in patients with extensive-stage small cell lung cancer who had achieved complete response, partial response, or stable disease with their previous platinum chemotherapy regimen, such as cisplatin or carboplatin in combination with etoposide or irinotecan. In addition, the safety and effectiveness of sunitinib will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed extensive-stage SCLC. Extensive-stage is defined as disease that extends beyond one hemithorax and regional lymph nodes (ipsilateral or contralateral hilar, mediastinal, or supraclavicular lymph nodes), or with cytologically positive pleural effusion.
* Patients who have completed platinum-based chemotherapy and demonstrated a complete response, partial response, or stable disease can be registered on the trial. A maximum of 4 cycles of induction chemotherapy is allowed. Patients must begin therapy within 28-42 days after day 1 of the 4th cycle of induction therapy and within 28 days of scans demonstrating stable disease or better. Prior palliative radiation therapy will be allowed as long as radiation was completed at least 1 week before starting protocol therapy.
* Resolution of all acute toxic effects of prior chemotherapy or radiotherapy or surgical procedures to NCI CTCAE Version 3.0 grade 1.
* Age * 18 years with Southwest Oncology Group (SWOG) performance status of 0,1 or 2 (Appendix 2).
* Adequate organ function as evidenced by the laboratory values listed in the protocol

Exclusion Criteria:

* Symptomatic or untreated brain or leptomeningeal metastases. Treated patients should be neurologically stable for at least 2 weeks after completion of appropriate therapy without the use of steroids. Patients currently on steroids are ineligible.
* More than 4 cycles of induction chemotherapy. Patients will be eligible for if they have completed at least 2 cycles of platinum-based induction chemotherapy and they have exhibited a complete or partial response to therapy. Patients who have received less than 4 cycles of induction chemotherapy and have less than a partial response will not be eligible.
* NCI CTCAE grade 3 hemorrhage within 4 weeks of starting the study treatment.
* History of gross hemoptysis due to lung cancer.
* Previous or concurrent malignancies, with the exception of adequately treated squamous cell or basal cell carcinoma of the skin, in situ carcinoma of the cervix, or any other malignancy treated and in clinical remission for more than 3 years.
* Major surgery or within 4 weeks of starting study treatment.
* Any history of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (CHF), cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
* Ongoing cardiac dysrhythmias
* Hypertension that cannot be controlled by medications
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication.
* Therapeutic anticoagulation with warfarin or heparin.
* Serious concomitant medical illness, including, but not limited to, uncontrolled angina, myocardial infarction and/or stroke within 3 months, or HIV infection.
* Acute or chronic liver disease
* History of dementia, active psychiatric disorder or any other condition, considered by the treating physician to impair the patient's ability to take oral pills on a daily basis or comply with the protocol requirements.
* Pregnant or lactating females.
* Use of agents with proarrhythmic potential is not permitted during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Kalemkerian, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Schneider BJ, Gadgeel SM, Ramnath N, Wozniak AJ, Dy GK, Daignault S, Kalemkerian GP. Phase II trial of sunitinib maintenance therapy after platinum-based chemotherapy in patients with extensive-stage small cell lung cancer. J Thorac Oncol. 2011 Jun;6(6):1117-20. doi: 10.1097/JTO.0b013e31821529c3. PMID 21512407

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16 subjects recruited from 7/19/2007 to 2/1/2010 at University of Michigan, Ann Arbor(lead site), and sub-sites: The University of Detroit's Karmanos Cancer Institute, WSU, Detroit; Weill Cornell Medical College, NY; and Roswell Park Cancer Institute, NJ
Pre-assignment Details: Patients with histologically or cytologically documented Extensive-Stage Small Cell Lung Cancer (ES-SCLC) who had received no more than 4 cycles of frontline platinum plus etoposide chemotherapy and who demonstrated a response or stable disease were eligible. ES-SCLC was defined as disease extending beyond 1 hemothorax and regional lymph nodes.
Groups:
- Sunitinib Maintenance Therapy: Sunitinib 50 mg po QD × 28 days followed by a 14 day break every 42 days until disease progression or unacceptable toxicity. Treatment to begin 28-42 days after day 1 of the last cycle of induction chemotherapy to allow confirmation of response or disease stability with chemotherapy.
Period: Overall Study
Arm/Group | Sunitinib Maintenance Therapy
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Lung cancer patients who are greater than or equal to 18 years old, who have had a response or maintained stable disease after undergoing no more that 4 cycles with platinum with etoposide chemotherapy
Arm/Group | Sunitinib Maintenance Therapy
Number analyzed (Participants) | 16
Age, Customized [Mean (Full Range); unit: years] | 66 [34 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 16
Response to induction chemotherapy [Number; unit: participants] — Per response evaluation criteria in Solid Tumors Criteria (RECIST v. 1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR) >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
  participants
    CR (complete response) | 3
    PR (partial response) | 11
    SD (stable disease) | 2
Performance status [Number; unit: participants] — The "Zubrod Performance Scale" is a measure of a lung cancer patient's functionality and condition. The measure ranks patients on a scale from 0-5, with 0 being fully active and asymptomatic, 1 being symptomatic but completely ambulatory, 2 being symptomatic and 50% in bed during day, 3 being symptomatic and more than 50% in bed, but not bedbound; 4 being bedbound or completely disabled; and 5 being moribund.
  participants
    0 | 5
    1 | 10
    2 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Rate
Description: The proportion of patients who are progression-free at 4 months after starting sunitinib.
Time Frame: 4 Months Post Treatment
Population: All 16 patients enrolled received a median of 4 weeks sunitinib maintenance therapy. 1 patient who discontinued requested no follow up and was censored from survival analysis. All survival endpoints were analyzed using the Kaplan-Meier method (Kaplan El, Meier P, Non-parametric Estimation from Incomplete Observations, J Am Stat Association, 1958)
Measure: Number (95% Confidence Interval); unit: percentage of patients with PFS
Groups:
- Sunitinib Maintenance Therapy: Sunitinib 50 mg po QD × 28 days followed by a 14 day break every 42 days until disease progression or unacceptable toxicity. Treatment to begin 28-42 days after day 1 of the last cycle of induction chemotherapy to allow confirmation of response or disease stability with chemotherapy. All patients who have received at least one cycle of sunitinib will be considered evaluable for response.
Arm/Group | Sunitinib Maintenance Therapy
Number analyzed (Participants) | 16
percentage of patients with PFS | 13 [2 to 33]

2. Secondary Outcome: Median Overall Survival
Description: Survival will be defined as the time from the first day of therapy to the date of death. If the patient is lost to follow-up, survival will be censored on the last date the patient was known to be alive. Survival for induction therapy will be calculated from day 1 of first cycle of chemotherapy. Survival for post-induction therapy will be calculated from the date the patient starts sunitinib.
Time Frame: up to 4 months post treatment
Population: 15 participants in Sunitinib maintenance therapy (main study) were enrolled and were evaluable for this outcome measure. Although 16 patients were enrolled, one patient opted to discontinue therapy, refused further follow-up, and was therefore censored from survival analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib Maintenance Therapy
Number analyzed (Participants) | 15
months | 8.2 [6.2 to 14.7]

3. Secondary Outcome: Percent of Patients With an Objective Response
Description: Scans were performed every 2 cycles to evaluate for response/progression. Response was assessed according to RECIST (Response Evaluation Criteria in Solid Tumors) criteria. Patients would be considered to have an objective response if they experience CR (Complete Response - Disappearance of all clinical and radiological evidence of target lesions and/or non-target lesions) or PR (Partial Response - A 30% or greater decrease in the sum of LD of all lesions in reference to the baseline sum LD).
Time Frame: 12 weeks (2 cycles)
Population: Patients who received at least 2 cycles of study therapy (maintenance sunitinib)
Measure: Number; unit: percentage of participants
Arm/Group | Sunitinib Maintenance Therapy
Number analyzed (Participants) | 15
percentage of participants | 0

4. Secondary Outcome: Number of Patients That Discontinue Drug Due to Toxicity
Description: Tolerability of Sunitinib will be evaluated by looking at the number of participants who discontinue drug due to toxicity. Toxicity was graded according to the National Cancer Institute (NCI) Common Toxicity Criteria v.3.0.
  In the event of any CTC, version 3.0 drug-related grade 3 or 4 non-hematologic or grade 4 hematologic adverse event(s), drug should be held until the toxicity resolves to < grade 1 and then the drug should be restarted at a one dose-level reduction.
  Recovery to acceptable levels of toxicity must occur within 4 weeks to allow continuation in the study.
  No more than 2 dose reductions are permitted for any patient. If further dose reduction is required, the patient must be removed from the study.
Time Frame: 20 weeks
Population: All patients who received sunitinib maintenance therapy were evaluable for toxicity and tolerability analysis.
Measure: Number; unit: participants
Arm/Group | Sunitinib Maintenance Therapy
Number analyzed (Participants) | 16
participants | 5

ADVERSE EVENTS:
Time Frame: Participants were evaluated for toxicity if they received sunitinib maintenance therapy (at least one dose) from onset of this therapy until the participant ended participation.
Description: Treatment was held for Participants with grade 4 hematologic or grade 3-4 non-hematologic toxicities until resolution to grade 2 or less. Treatment was then restarted at a dose of 3.75 mg. A second dose reduction to 25 mg was permitted. Treatment discontinued for a third dose reduction or life-threatening, irreversible or unacceptable toxicity.
Arm/Group | Sunitinib Maintenance Therapy
Serious Adverse Events (participants affected / at risk) | 4/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib Maintenance Therapy (N=16)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 (1)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 1 (1)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Death (General disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (2)
Infection, Lung (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain in extremity (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib Maintenance Therapy (N=16)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Ataxia (Nervous system disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Decubitus (Skin and subcutaneous tissue disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 5 (7)
Dyspepsia (Gastrointestinal disorders) | 3 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Edema limbs (General disorders) | 2 (3)
Fatigue (General disorders) | 10 (15)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 6 (6)
Hemoglobin (Blood and lymphatic system disorders) | 3 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Leukocytes (Blood and lymphatic system disorders) | 5 (6)
Mucositis oral (Gastrointestinal disorders) | 3 (6)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 10 (12)
Neutrophils (Blood and lymphatic system disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Platelet count decreased (Blood and lymphatic system disorders) | 2 (3)
Platelets (Blood and lymphatic system disorders) | 7 (11)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (3)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (2)
Speech disorder (Nervous system disorders) | 2 (3)
Sweating (Skin and subcutaneous tissue disorders) | 2 (2)
Taste alteration (Gastrointestinal disorders) | 3 (3)
Urine discoloration (Renal and urinary disorders) | 3 (3)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 7 (7)
Weight loss (Investigations) | 4 (6)

LIMITATIONS AND CAVEATS:
The trial was to be terminated at stage 1 if less than, or equal to, 8 patients were progression free at 4 months. The PFS rate did not reach the threshold required for study continuation and, therefore, the study was discontinued early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No